CLINICAL TRIAL: NCT04887571
Title: the PrEsentation, Rationale and Impact of reperFUSION for Acute Coronary Syndromes in Cape Town and the Garden Route Health District - the PERFUSION Registry
Acronym: PERFUSION
Status: Completed | Type: Observational
Sponsor: University of Cape Town (Other)
Responsible Party: Principal Investigator, Kishal Lukhna, Dr, University of Cape Town
Other Study IDs: PERFUSION
Record Dates: First submitted 2021-05-05; First posted 2021-05-14 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Acute Coronary Syndrome; ST Elevated Myocardial Infarction; Non ST Elevation Myocardial Infarction; Unstable Angina
Keywords: Acute Coronary Syndrome; STEMI; NSTEMI; Unstable Angina; Sub-Saharan Africa; Cape Town; South Africa; Myocardial Infarction
MeSH Terms: conditions — Acute Coronary Syndrome; ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction; Angina, Unstable; Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational ACS Registry: All consecutive adult patients in the Cape Metropole and the Garden Route Health District with an acute coronary syndrome will be recruited into the PERFUSION registry across the study duration.
  Interventions: Other: No Intervention - Observational Registry

INTERVENTIONS:
Other: No Intervention - Observational Registry — All consecutive adult patients in the Cape Metropole and the Garden Route Health District with an Acute coronary syndrome (STEMI, NSTEMI, Unstable Angina) will be recruited into the PERFUSION Registry.

SUMMARY:
The global burden and threat of non-communicable diseases (NCDs) have become a major health challenge that undermines social and economic development throughout the world. Cardiovascular disease including acute coronary syndromes (ACS) currently accounts for 17.9 million deaths a year. Low and middle-income countries such as those in sub-Saharan Africa (SSA) have undergone a rapid epidemiological transition over the last few decades and now have a burden of disease increasingly dominated by NCDs. The global burden of disease report for 2017 revealed a 71.4% increase in cardiovascular disease in SSA, predicting a large increase in mortality. Unfortunately, reliable population-level data regarding the incidence, prevalence and demographics of ACS in SSA are limited. The investigators propose to set up and conduct a multi-centre, prospective, observational registry to describe the demographics, clinical characteristics, presentation, management and outcomes of patients admitted with ACS in Cape Town and the Garden Route Health District, Western Cape Province, South Africa. The registry is designed to shed insight on the current burden and impact of atherosclerotic cardiovascular disease in the Western Cape.

DETAILED DESCRIPTION:
The investigators propose to set up and conduct a multi-centre, prospective, observational registry to describe the demographics, clinical characteristics, presentation, management and outcomes of patients admitted with ACS in Cape Town and the Garden Route Health District, Western Cape Province, South Africa.

The aims of this prospective multi-centre registry are to describe the burden, demographics, risk factor profile, clinical course, management, and outcomes of patients presenting with ACS across the Cape Town metropole and the Garden Route Health District. The registry will be called "the PrEsentation, Rationale and impact of reperFUSION for Acute Coronary Syndromes in Cape Town - the PERFUSION registry". It will be designed to determine the feasibility of conducting a large multi-centre Acute Coronary Syndrome registry in South Africa.

Primary Objectives:

1. to enrol consecutive patients presenting with acute coronary syndromes from designated participating sites;
2. to describe the demographic and risk factor profile of participants with ACS;
3. to describe the burden of patients presenting with ACS in the Cape Town metropole and the Garden Route Health District;
4. to describe the management of patients with ACS and assess compliance with current South African guidelines;
5. to describe the one month, six-month and 12-month outcomes with regard to all-cause mortality, hospitalisation, and major adverse cardiac events (recurrence of ACS, heart failure, stroke and ventricular tachy-arrythmias).

Methods:

Registry design The PERFUSION registry will enrol consecutive consenting adults (≥ 18 years) admitted to participating healthcare centres in the cities of Cape Town and the Garden Route Health District, Western Cape, South Africa. Depending on available capacity and resources, the registry may be expanded to other healthcare centres in the Western Cape and other provinces of South Africa.

As this is fundamentally an observational study, all participants enrolled will receive management based on local standard of care guidelines. Participant management will not be affected by recruitment into this study. By using the hub/ spoke/ pre-spoke model, all patients presenting with an ACS to a designated public healthcare care facility in the Cape Town metropole and the Garden Route Health District will be screened for study eligibility criteria. Screening will occur at hub and spoke levels only. Designated site PI's will identify potential study participants meeting eligibility criteria during their index ACS admission. Once screened according to the study's inclusion and exclusion criteria, potential participants will be consented for study participation. Clinical information fulfilling pre-defined registry variables will be entered into a standardised paper-based case report form (CRF) or electronic CFR and uploaded onto a secure data collection web application called the Research Electronic Data Capture (REDCap) by the study's data capturers. Upon data entry, participants will be immediately assigned a unique identifier generated by REDCap to maintain confidentiality. The REDCap database is governed by strict password-controlled access, assigned only to approved study team members.

Data collection:

The database variables collected for this registry are in line with the American College of Cardiology Foundation / American Heart Association Task Force on Key Data Elements. These include data pertaining to patient demographics; comorbidities and prior medication; index ACS presentation at the pre-spoke, spoke or hub level; ECG features; echocardiography; laboratory investigations; management and treatment received at the pre-spoke, spoke or hub level; angiography; complications of therapies and interventions; and outcomes (in-hospital, 1 month, 6 month and 1 year).

To limit an additional burden on the healthcare system, the investigators plan on following-up participants electronically using the Western Cape Provincial Health Data Centre (PHDC) and Single Patient Viewer (SPV) online tool over a period of 1-year after the index ACS presentation. The investigators have received both HREC and provincial permission for the utilisation of data from the PHDC and SPV for this research. Follow-up data will be uploaded directly onto REDCap and anonymised.

The key outcomes of interest will include:

1. mortality (all-cause and cardiovascular);
2. recurrent and re-infarction myocardial infarction;
3. new-onset heart failure and arrhythmia complications;
4. cerebrovascular events;
5. major bleeding events;
6. repeat hospitalisation for any cause.

The extended list of all variables collected will be found on the registry's CRF.

Benefits of registry participation:

Although there are no direct study benefits to the participant, the study will indirectly improve our knowledge of acute coronary syndromes in South Africa. By providing local reliable evidence in our resource constraint environment, the investigators may improve the standard of care provided to patients with ACS and possibly identify novel cardioprotective strategies that may help reduce the burden of ACS in South Africa.

Risk of registry participation:

The PERFUSION registry is designed to be a prospective, observational registry. Participant enrolment will not deviate management from local standard of care guidelines. There is no investigational medicinal product, drug or device practised in this protocol. Participation in this study has no physical, psychological, social, economic or legal risk. For people who do not want to take part in the study, routine standard of care will be maintained.

ELIGIBILITY:
Inclusion Criteria:

* signed written informed consent before any study recruitment; and
* male or female patients age ≥ 18 years of age; and
* a diagnosis of ACS (STEMI, NSTEMI or UA).

Exclusion Criteria:

* ACS absent within index admission; or
* refusal of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study is designed to include adult patients from the Cape Metropole and the Garden Route Health District who present with acute coronary syndromes (STEMI, NSTEMI, or Unstable Angina).
Sampling Method: Non-Probability Sample
Enrollment: 870 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
1-year combined primary endpoint | 1 year
  all-cause death, cardiac death, re-hospitalisation myocardial infarction, cerebrovascular accident

SECONDARY OUTCOMES:
cardiac adverse events | 1-year
  re-hospitalisation for heart failure, or arrhythmias
1 month combined end point | 1-month
  all-cause death, cardiac death, re-hospitalisation myocardial infarction, cerebrovascular accident
6 month combined end point | 6-month
  all-cause death, cardiac death, re-hospitalisation myocardial infarction, cerebrovascular accident
Compliance profile | 1-year
  1-year compliance on guideline directed medical treatment
Refusion time | 1-year
  Time to ECG and reperfusion in patients with Acute Coronary Syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Mpiko Ntsekhe, PhD, Principal Investigator — Groote Schuur Hospital
Locations (4):
- South Africa (4):
  - Groote Schuur Hospital, Cape Town, Western Cape
  - Victoria Hospital, Cape Town, Western Cape
  - New Somerset Hospital, Cape Town, Western Cape
  - George Hospital, George, Western Cape

IPD SHARING:
Plan to Share IPD: Undecided